CLINICAL TRIAL: NCT05067452
Title: Pilot Study of the Nutrition-Supported Diabetes Education Program (NU-DSMP) Among Low-Income Adults With Type 2 Diabetes
Brief Title: Pilot Trial of the Nutrition-Supported Diabetes Education Program
Acronym: NU-DSMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Project Open Hand (Other); Contra Costa Health Services (Other Government); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: R21DK123632 (NIH); R21DK123632 (NIH)
Record Dates: First submitted 2021-09-21; First posted 2021-10-05 (Actual); Results first posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: food security; nutrition
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Case Management

STUDY DESIGN:
Intervention Model Description: Participants (n=72) will be randomized to the intervention (n=36) or control (n=36) arms. The intervention consists of providing diabetes-tailored food support and individualized case management over 12 weeks to patients with type 2 diabetes.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The analyst(s) and investigator(s) conducting and reviewing the analyses of the data will be masked to whether participants were in the intervention or control arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care including diabetes self-management education (No Intervention): Control participants will receive standard of care as offered by clinical partners to all T2DM patients, including referral to nutritional counseling, T2DM support groups, and participation in local diabetes self-management programs. Control participants are also often provided referral information for locally available food support services in the region that provide diabetes-appropriate foods. Control participants will participate in the Diabetes Self-Management Program, an evidence-based program that takes place over 6 weeks that meets the standard of care for diabetes education.
  At the end of follow up, the control arm will receive three months diabetes-tailored food support consisting of diabetes-tailored grocery boxes and nutrition case-management.
- Diabetes-tailored food support plus diabetes self-management education (Experimental): The intervention has two components: 1) diabetes-tailored food support that consists of weekly, home-delivered medically tailored meals, and monthly home-delivered healthy groceries, from baseline to 24 weeks, and 2) three case-management sessions with client services staff from the partnering nutrition agency over the 12 weeks of intervention.
  The intervention will be delivered in addition to a base condition consisting of remote participation in the Diabetes Self-Management Program, an evidence-based diabetes education program that takes place over 6 weeks also received by the control group as part of the standard of care.
  Interventions: Other: Food support; Other: Case-management

INTERVENTIONS:
Other: Food support — Diabetes-tailored food support. Project Open Hand (POH) will provide intervention participants twelve weeks of supplemental food support. Food support will consist of a mix of meals tailored for T2DM, and T2DM-healthy groceries, consistent with American Diabetes Association (ADA) guidelines for diabetes healthy diets under the responsibility of a registered dietitian. All food support will be home delivered.
  Arms: Diabetes-tailored food support plus diabetes self-management education
Other: Case-management — Project Open Hand client services staff will conduct three case management sessions with the participant. The first session will initiate food services and ensure orientation to the intervention and set up delivery; the second session will support the participant with any issues related to the intervention (logistical or nutrition-related, with referral to the POH registered dietitian as needed); the third session will provide transition from the intervention, connect the participant with local food resources, and ensure a "warm hand-off" to nutrition
  Arms: Diabetes-tailored food support plus diabetes self-management education

SUMMARY:
This is a pragmatic, pilot randomized controlled trial (RCT) of the Nutrition-Supported Diabetes Education Program (NU-DSMP). This study will test the feasibility and preliminary impact of providing diabetes-tailored food support and individualized case-management on glycemic control and other intermediate outcomes including food security, diet, mental health, and health care behaviors, among Medicaid-enrolled patients with type 2 diabetes in a safety-net county health system.

DETAILED DESCRIPTION:
Together with Contra Costa Health Services, a safety-net county health system, and Project Open Hand, a non-profit organization with extensive experience providing nutrition services to low-income, chronically ill individuals in the San Francisco Bay Area, the investigators will conduct the Nutrition-Supported Diabetes Education Program (NU-DSMP) Pilot Study. The goal for this pragmatic, pilot randomized trial is to test the feasibility, acceptability and preliminary impact of providing 12 weeks of diabetes-healthy food support (i.e. medically tailored meals and groceries) supported by individualized case-management to low-income individuals with type 2 diabetes mellitus (T2DM) participating in the evidence-based Diabetes Self- Management Program (DSMP), compared to DSMP participation alone.

The study will randomize 72 individuals 1:1 to intervention and control arms, following them at 0, 12 and 24 weeks with surveys and medical record review (with an interim brief 6 week assessment with the survey only), to understand the impact on diabetes health. Data from this pilot study will inform the planning of a full-size randomized trial to test the efficacy of the NU-DSMP model, with a long-term goal to inform policy debates about the value of implementing medically tailored food interventions as part of healthcare.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of type 2 diabetes mellitus (T2DM) in the medical record
* Most recent HbA1c (within 1 year) ≥ 7%
* Receives primary care for diabetes from Contra Costa Health Services
* Is a current member of Contra Costa Health Plan
* Age ≥18 years
* Has an HbA1c test in the medical record in the last month; OR their doctor has an active order for an HbA1c test for the potential participant; OR the participant is eligible to have a test ordered as part of usual care
* Speaks English or Spanish
* Adequate cognitive and hearing capacity to complete study measures
* Willing to participate in the online or telephone DSMP education, and if randomized to the intervention, to receive home-delivered meals and groceries
* Has the ability to engage with simple reading materials (e.g. directions to join the education session by phone or Zoom) on their own or with the support of a family member or friend
* Has access to a device (telephone, tablet, and/or computer) that can be used to receive remote DSMP education (possible via phone, computer or tablet) and complete study assessments (phone only; or tablet or computer with phone capabilities) (does not need to be participant's own device)

Exclusion Criteria:

* Currently pregnant at baseline, currently breastfeeding, up to 6 months postpartum, or plans to become pregnant during the course of the study. If participant becomes pregnant during the study, services provided as part of the study won't stop, however, data will not be used in the main analysis
* Has confirmed Type 1 DM
* Has confirmed stage 5 chronic kidney disease, end stage renal disease or is on dialysis or expected to start dialysis in the next 6 months
* Does not have access to facilities to receive delivery of, store, and heat or prepare intervention food
* Has a food allergy, intolerance or preferred diet that POH cannot accommodate with meal delivery (e.g. vegan diet). POH can accommodate many but not all diet restrictions.
* Does not live in Contra Costa County or plans to move out of the county in the next 6 months
* Another household member is already enrolled in the NU-DSMP study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2023-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kartika Palar, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Contra Costa Health Services, Martinez, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care and Diabetes Self-management Education: Control participants will receive standard of care as offered by clinical partners to all type 2 diabetes mellitus (T2DM) patients, including referral to nutritional counseling, T2DM support groups, and participation in local diabetes self-management programs. Control participants are also often provided referral information for locally available food support services in the region that provide diabetes-appropriate foods. Control participants will participate in the Diabetes Self-Management Program, an evidence-based program that takes place over 6 weeks that meets the standard of care for diabetes education.
  At the end of follow up, the control arm will receive three months diabetes-tailored food support consisting of diabetes-tailored grocery boxes and nutrition case-management.
- Diabetes-tailored Food Support Plus Diabetes Self-management Education: The intervention has two components: 1) diabetes-tailored food support that consists of weekly, home-delivered medically tailored meals, and monthly home-delivered healthy groceries, from baseline to 24 weeks, and 2) three case-management sessions with client services staff from the partnering nutrition agency over the 12 weeks of intervention.
  The intervention will be delivered in addition to a base condition consisting of remote participation in the Diabetes Self-Management Program, an evidence-based diabetes education program that takes place over 6 weeks (same as control group).
  Food support: Diabetes-tailored food support. Project Open Hand (POH) will provide intervention participants twelve weeks of supplemental food support. Food support will consist of a mix of meals tailored for T2DM, and T2DM-healthy groceries, consistent with American Diabetes Association (ADA) guidelines for diabetes healthy diets under the responsibility of a registered dietitian. All food support will be home delivered.
  Case-management: Project Open Hand client services staff will conduct three case management sessions with the participant. The first session will initiate food services and ensure orientation to the intervention and set up delivery; the second session will support the participant with any issues related to the intervention; the third session will provide transition from the intervention and connect the participant with local food resources.
Period: Overall Study
Arm/Group | Standard of Care and Diabetes Self-management Education | Diabetes-tailored Food Support Plus Diabetes Self-management Education
Started | 15 | 21
Completed | 15 | 17
Not Completed | 0 | 4
Not completed — Lost to Follow-up | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Standard of Care and Diabetes Self-management Education: Control participants will receive standard of care as offered by clinical partners to all T2DM patients, including referral to nutritional counseling, T2DM support groups, and participation in local diabetes self-management programs. Control participants are also often provided referral information for locally available food support services in the region that provide diabetes-appropriate foods. Control participants will participate in the Diabetes Self-Management Program, an evidence-based program that takes place over 6 weeks that meets the standard of care for diabetes education.
  At the end of follow up, the control arm will receive three months diabetes-tailored food support consisting of diabetes-tailored grocery boxes and nutrition case-management.
- Diabetes-tailored Food Support Plus Diabetes Self-management Education: The intervention has two components: 1) diabetes-tailored food support that consists of weekly, home-delivered medically tailored meals, and monthly home-delivered healthy groceries, from baseline to 24 weeks, and 2) three case-management sessions with client services staff from the partnering nutrition agency over the 12 weeks of intervention.
  The intervention will be delivered in addition to a base condition consisting of remote participation in the Diabetes Self-Management Program, an evidence-based diabetes education program that takes place over 6 weeks (same as control group).
  Food support: Diabetes-tailored food support. Project Open Hand will provide intervention participants twelve weeks of supplemental food support. Food support will consist of a mix of meals tailored for T2DM, and T2DM-healthy groceries, consistent with American Diabetes Association (ADA) guidelines for diabetes healthy diets under the responsibility of a registered dietitian. All food support will be home delivered.
  Case-management: Project Open Hand client services staff will conduct three case management sessions with the participant. The first session will initiate food services and ensure orientation to the intervention and set up delivery; the second session will support the participant with any issues related to the intervention; the third session will provide transition from the intervention and connect the participant with local food resources.
- Total: Total of all reporting groups
Arm/Group | Standard of Care and Diabetes Self-management Education | Diabetes-tailored Food Support Plus Diabetes Self-management Education | Total
Number analyzed (Participants) | 15 | 21 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (10.6) | 56.0 (12.6) | 54.1 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 28
  Male | 2 | 6 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White, Caucasian | 0 | 3 | 3
  Race/Ethnicity: Black, African American | 4 | 4 | 8
  Race/Ethnicity: Hispanic, Latino | 11 | 11 | 22
  Race/Ethnicity: Asian, Pacific Islander | 0 | 1 | 1
  Race/Ethnicity: American Indian, Native American | 0 | 0 | 0
  Race/Ethnicity: Other race/ethnicity | 0 | 1 | 1
  Race/Ethnicity: More than one race/ethnicity | 0 | 1 | 1
Education [Count of Participants; unit: Participants]
  Less than high school | 8 | 6 | 14
  High school/GED | 5 | 4 | 9
  More than high school | 2 | 11 | 13
Annual household income [Count of Participants; unit: Participants]
  Less than $10,000 | 6 | 6 | 12
  $10,000 to $20,000 | 4 | 12 | 16
  $20,000 to $30,000 | 4 | 0 | 4
  $30,000 to $40,000 | 0 | 1 | 1
  Over $40,000 | 0 | 2 | 2
  Refused to answer | 1 | 0 | 1
Has child dependents [Count of Participants; unit: Participants] | 8 | 8 | 16
HbA1c (%) [Mean (Standard Deviation); unit: Percentage of glycated hemoglobin] — Population: Error in laboratory result; one baseline value implausibly high (30.5). The value was removed (intervention group).
  Percentage of glycated hemoglobin
    number analyzed (Participants) | 15 | 20 | 35
    (all) | 8.69 (1.70) | 8.24 (1.68) | 8.43 (1.68)
HbA1c < 9% [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description: Error in laboratory result; one baseline value implausibly high (30.5). The value was removed (intervention group).
  Participants
    number analyzed (Participants) | 15 | 20 | 35
    (all) | 9 | 15 | 24
Food security score [Mean (Standard Deviation); unit: units on a scale] — USDA Household Food Security Survey Module - 10 item (adult items). The score ranges from 0 to 10. A higher score indicates a higher severity of food insecurity.
  units on a scale | 3.20 (2.83) | 3.00 (2.83) | 3.08 (2.79)
Low or very low food security [Count of Participants; unit: Participants] — USDA Household Food Security Survey Module - 10 item (adult items)
  Participants | 8 | 11 | 19
Healthy days (last 30 days) [Mean (Standard Deviation); unit: days] | 16.2 (13.3) | 13.3 (13.3) | 14.5 (13.2)
Fruit and vegetable consumption [Mean (Standard Deviation); unit: Cup equivalents per day] | 2.53 (1.19) | 2.60 (1.03) | 2.57 (0.987)
Added sugar consumption [Mean (Standard Deviation); unit: teaspoon equivalents per day] | 11.94 (2.45) | 12.4 (2.52) | 12.2 (2.46)
Depressive symptom severity score (PHQ-8) [Mean (Standard Deviation); unit: units on a scale] — The PHQ-8 score ranges from 0 to 24, with higher scores indicating higher severity of depressive symptoms.
  units on a scale | 5.13 (6.32) | 8.05 (6.21) | 6.83 (6.34)
Diabetes self-efficacy score [Mean (Standard Deviation); unit: units on a scale] — The 8-item Diabetes Self-Efficacy scale was used to assess confidence in one's ability to manage numerous self-care behaviors. Scores range from 8 to 40, with higher scores indicating more confidence in self-managing their diabetes.
  units on a scale | 29.2 (4.71) | 30.5 (4.35) | 30.0 (4.49)

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin A1c (HbA1c) From Baseline to Twelve Weeks by Study Arm
Description: Change HbA1c levels (%) from baseline to twelve weeks by study arms
Time Frame: Baseline and twelve weeks
Measure: Mean (Standard Deviation); unit: Percentage of glycated hemoglobin
Arm/Group | Standard of Care and Diabetes Self-management Education | Diabetes-tailored Food Support Plus Diabetes Self-management Education
Number analyzed (Participants) | 13 | 13
Percentage of glycated hemoglobin | -0.023 (1.63) | 0.131 (2.14)
Statistical Analysis 1: Comparison: Standard of Care and Diabetes Self-management Education vs Diabetes-tailored Food Support Plus Diabetes Self-management Education; Test type: Superiority; p = 0.900, ANCOVA; Slope = -0.092, 95% CI 2-sided [-1.59 to 1.40], Standard Error of Mean 0.721

2. Primary Outcome: Change in Food Security Severity From Baseline to Twelve Weeks by Study Arm
Description: The US household food security survey module (adult version) from the US Department of Agriculture (USDA) will be used to assess the change in the food security scores from baseline to twelve weeks. The score ranges from 0 to 10. Higher score indicates higher severity of food insecurity.
Time Frame: Baseline and twelve weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard of Care and Diabetes Self-management Education | Diabetes-tailored Food Support Plus Diabetes Self-management Education
Number analyzed (Participants) | 13 | 15
score on a scale | -1.31 (3.17) | 0.067 (1.71)
Statistical Analysis 1: Comparison: Standard of Care and Diabetes Self-management Education vs Diabetes-tailored Food Support Plus Diabetes Self-management Education; Test type: Superiority; p = 0.146, Mixed Models Analysis; Slope = 1.37, 95% CI 2-sided [-0.478 to 3.23], Standard Error of Mean 0.945

3. Secondary Outcome: Change in the Percentage of Participants With Glucose Control From Baseline to Twelve Weeks by Study Arm
Description: Glucose control will be defined as HbA1c lower than 9%. The change from baseline to twelve weeks, in the percentage of participants with glucose control will be reported.
Time Frame: Baseline and twelve weeks
Measure: Number; unit: Percentage of participants
Arm/Group | Standard of Care and Diabetes Self-management Education | Diabetes-tailored Food Support Plus Diabetes Self-management Education
Number analyzed (Participants) | 13 | 13
Percentage of participants | 7.70 | -7.70
Statistical Analysis 1: Comparison: Standard of Care and Diabetes Self-management Education vs Diabetes-tailored Food Support Plus Diabetes Self-management Education; Test type: Superiority; p = 0.281, ANCOVA; Linear regression used with the binary outcome (linear probability model); Risk Difference (RD) = 0.235, 95% CI 2-sided [-0.207 to 0.677], Standard Error of Mean 0.212

4. Secondary Outcome: Change in the Percentage of Participants With Low and Very Low Food Security From Baseline to Twelve Weeks by Study Arm
Description: Low and very low food security will be defined as 3 or more items answered affirmatively in the USDA's US household food security survey module. Change in the percentage of participants with low or very low food security, from baseline to twelve weeks by intervention arms will be reported.
Time Frame: Baseline and twelve weeks
Measure: Number; unit: Percentage of participants
Arm/Group | Standard of Care and Diabetes Self-management Education | Diabetes-tailored Food Support Plus Diabetes Self-management Education
Number analyzed (Participants) | 13 | 15
Percentage of participants | -15.4 | 20
Statistical Analysis 1: Comparison: Standard of Care and Diabetes Self-management Education vs Diabetes-tailored Food Support Plus Diabetes Self-management Education; Test type: Superiority; p = 0.094, Mixed Models Analysis; Linear regression used with the binary outcome (linear probability model); Risk Difference (RD) = 0.354, 95% CI 2-sided [-0.060 to 0.768], Standard Error of Mean 0.211

5. Secondary Outcome: Change in Health-related Quality of Life (Healthy Days) From Baseline to Twelve Weeks by Study Arm
Description: Health-related quality of life will be measured using the Summary Index of Unhealthy Days collected via the Centers for Disease Control (CDC) Healthy Days scale. This scale asks the number of days in the past 30 days the person felt physically or mentally unwell. The summary index then estimates the number of recent days when a person's physical and mental health was good (or better) and is calculated by subtracting the number of unhealthy days from 30 days. The change in healthy days from baseline to twelve weeks by study arm will be reported.
Time Frame: Baseline and twelve weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Standard of Care and Diabetes Self-management Education | Diabetes-tailored Food Support Plus Diabetes Self-management Education
Number analyzed (Participants) | 13 | 15
days | -1.38 (9.39) | 0.800 (16.2)
Statistical Analysis 1: Comparison: Standard of Care and Diabetes Self-management Education vs Diabetes-tailored Food Support Plus Diabetes Self-management Education; Test type: Superiority; p = 0.669, Mixed Models Analysis; Slope = 2.18, 95% CI 2-sided [-7.83 to 12.2], Standard Error of Mean 5.11

6. Secondary Outcome: Change in Consumption of Fruits and Vegetables From Baseline to Twelve Weeks by Study Arm
Description: Dietary information using the Dietary Screener Questionnaire (DSQ) will be collected. The DSQ obtains information on the frequency of consumption of fruits and vegetables. These responses are then converted to cup equivalents per day using a scoring algorithm based on the NHANES 24-hour recall. Fruit and vegetable consumption from baseline to twelve weeks by study arm will be reported.
Time Frame: Baseline and twelve weeks
Measure: Mean (Standard Deviation); unit: cup equivalents
Arm/Group | Standard of Care and Diabetes Self-management Education | Diabetes-tailored Food Support Plus Diabetes Self-management Education
Number analyzed (Participants) | 13 | 15
cup equivalents | 0.294 (0.962) | 0.317 (0.973)
Statistical Analysis 1: Comparison: Standard of Care and Diabetes Self-management Education vs Diabetes-tailored Food Support Plus Diabetes Self-management Education; Test type: Superiority; p = 0.949, Mixed Models Analysis; Slope = -0.024, 95% CI 2-sided [-0.695 to 0.743], Standard Error of Mean 0.367

7. Secondary Outcome: Change in Consumption of Added Sugars From Baseline to Twelve Weeks by Study Arm
Description: Dietary information using the Dietary Screener Questionnaire (DSQ) will be collected. The DSQ obtains information on the frequency of consumption of added sugars. These responses are then converted to teaspoon equivalents per day using a scoring algorithm based on the NHANES 24-hour recall. Added sugars consumption (teaspoon equivalents per day) from baseline to twelve weeks by study arm will be reported.
Time Frame: Baseline and twelve weeks
Measure: Mean (Standard Deviation); unit: teaspoon equivalents
Arm/Group | Standard of Care and Diabetes Self-management Education | Diabetes-tailored Food Support Plus Diabetes Self-management Education
Number analyzed (Participants) | 13 | 15
teaspoon equivalents | -0.405 (0.871) | -0.944 (1.73)
Statistical Analysis 1: Comparison: Standard of Care and Diabetes Self-management Education vs Diabetes-tailored Food Support Plus Diabetes Self-management Education; Test type: Superiority; p = 0.308, Mixed Models Analysis; Slope = -0.540, 95% CI 2-sided [-1.58 to 0.679], Standard Error of Mean 0.530

8. Secondary Outcome: Change in Depressive Symptoms From Baseline to Twelve Weeks by Study Arm
Description: The 8-item Patient Health Questionnaire (PHQ-8) will be used to evaluate depressive symptoms. The PHQ-8 score ranges from 0 to 24, with higher scores indicating higher levels of depression. The change in PHQ-8 scores from baseline to twelve weeks by study arm will be reported.
Time Frame: Baseline and twelve weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard of Care and Diabetes Self-management Education | Diabetes-tailored Food Support Plus Diabetes Self-management Education
Number analyzed (Participants) | 13 | 15
score on a scale | 0.154 (2.70) | -0.867 (6.40)
Statistical Analysis 1: Comparison: Standard of Care and Diabetes Self-management Education vs Diabetes-tailored Food Support Plus Diabetes Self-management Education; Test type: Superiority; p = 0.593, Mixed Models Analysis; Slope = -1.02, 95% CI 2-sided [-4.77 to 0.499], Standard Error of Mean 1.91

9. Secondary Outcome: Change in Diabetes Self-efficacy From Baseline to Twelve Weeks by Study Arm
Description: The 8-item Diabetes Self-Efficacy scale will be used to assess confidence in one's ability to manage numerous self-care behaviors. The scores ranges from 8 to 40, with higher scores indicating more confidence in self-managing their diabetes. The changes in the scores from baseline to twelve weeks by study arm will be reported.
Time Frame: Baseline and twelve weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard of Care and Diabetes Self-management Education | Diabetes-tailored Food Support Plus Diabetes Self-management Education
Number analyzed (Participants) | 13 | 15
score on a scale | 2.69 (3.84) | 0.067 (4.76)
Statistical Analysis 1: Comparison: Standard of Care and Diabetes Self-management Education vs Diabetes-tailored Food Support Plus Diabetes Self-management Education; Test type: Superiority; p = 0.112, Mixed Models Analysis; Slope = -2.63, 95% CI 2-sided [-5.86 to 0.611], Standard Error of Mean 1.65

10. Other Pre Specified Outcome: Change in HbA1c Values From Twelve Weeks to Twenty-four Weeks by Study Arm
Description: To evaluate durability of changes, if any, in HbA1c after the intervention ended, the change in HbA1c levels (%) from 12 weeks to 24 weeks by study arm will be reported.
Time Frame: Twelve weeks and twenty-four weeks
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Change in the Proportion of Participants With Glycemic Control From Twelve Weeks to Twenty-four by Study Arm
Description: To evaluate durability of changes, if any, in glycemic control after the intervention ended, the change in the percent of participants with HbA1c levels less than 9% from 12 weeks to 24 weeks by study arm will be reported.
Time Frame: Twelve weeks and twenty-four weeks
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Change in Health-related Quality of Life (Healthy Days) From Twelve Weeks to Twenty-four Weeks by Study Arm
Description: Health-related quality of life will be measured using the Summary Index of Unhealthy Days collected via the CDC Healthy Days scale. This scale asks the number of days in the past 30 days the person felt physically or mentally unwell. The summary index then estimates the number of recent days when a person's physical and mental health was good (or better) and is calculated by subtracting the number of unhealthy days from 30 days. To evaluate the durability of changes, if any, in health-related quality of life, the change in healthy days from 12 weeks to 24 weeks by study arm will be reported.
Time Frame: Twelve weeks and twenty-four weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Standard of Care and Diabetes Self-management Education | Diabetes-tailored Food Support Plus Diabetes Self-management Education
Number analyzed (Participants) | 15 | 16
days | 1.31 (7.17) | -1.36 (7.59)
Statistical Analysis 1: Comparison: Standard of Care and Diabetes Self-management Education vs Diabetes-tailored Food Support Plus Diabetes Self-management Education; Test type: Superiority; p = 0.349, Mixed Models Analysis; Slope = -2.66, 95% CI 2-sided [-8.25 to 2.92], Standard Error of Mean 2.85

ADVERSE EVENTS:
Time Frame: Baseline to 24 months
Arm/Group | Standard of Care and Diabetes Self-management Education | Diabetes-tailored Food Support Plus Diabetes Self-management Education
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/21
Other Adverse Events (participants affected / at risk) | 0/15 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-17): https://cdn.clinicaltrials.gov/large-docs/52/NCT05067452/Prot_SAP_001.pdf